CLINICAL TRIAL: NCT06238505
Title: Acute Efficacy of Exercises Applied With Xbox and Biodex Devices in Pes Planus"
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, hazal genc, Principal Investigator, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023-19/02
Record Dates: First submitted 2024-01-26; First posted 2024-02-02 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-02

CONDITIONS: Pes Planus
Keywords: pes planus; exercise
MeSH Terms: conditions — Flatfoot; Motor Activity | interventions — Cadaverine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual (Experimental)
  Interventions: Other: Virtual
- biodex (Experimental)
  Interventions: Other: biodex

INTERVENTIONS:
Other: Virtual — application will be made with virtual reality device
  Arms: Virtual
Other: biodex — application will be made with biodex device
  Arms: biodex

SUMMARY:
.Pes planus; It can be defined as the valgus of the hindfoot while loading the foot, the disappearance of the medial longitudinal arch in the midfoot, and the supination of the forefoot relative to the hindfoot. It may also occur due to the fact that the medial longitudinal arch in the foot is lower than the required height according to the anatomical position. The parts of the foot that touch the ground are anatomically healthy in a person; They are the heads of the calcaneus tuberositas calcanei on the back of the foot and the 5 metatarsal bones on the front of the foot. In the standing position, 25% of our body weight is on the tuber calcanei, while 25% is on the 5 metatarsal bones. In individuals with pes planus, convergence of the sole of the midfoot to the ground may even result in the sole of the midfoot touching the ground at its advanced levels. It is one of the common foot deformities.

DETAILED DESCRIPTION:
pes planus can cause symptoms and dysfunction that are symptomatic or severe enough to limit patients' quality of life. Degeneration of the posterior tibial tendon may occur due to trauma, neuroarthropathy, neuromuscular disease and inflammatory arthritis. Among these, the most common cause of pes planus is the degeneration of the posterior tibial tendon.

The highest arch of the foot, the medical longitudinal arch calcaneus, talus, navicular, cuneiform and 1-2-3. It is formed by metatarsals. It is effective in the distribution of the load on the feet. Plantar ligaments are important in protecting the dome of the foot.

They used many definitions known as pes planus, that is, flat feet in the literature. Weak foot, relaxed foot, pes valgus, congenital hypermobile flat foot, hypermobile flat foot, flaccid flat food, talipes calcaneovalgus, compensated talipes equinus can be given as examples.

ELIGIBILITY:
Inclusion Criteria:

* Having mild and moderate pes planus,
* Volunteering of individuals,
* Being between the age group of 18-25,
* Having experienced at least one inflammatory symptom (pain, swelling, etc.)
* Not having any systemic, locomotor and foot related diseases, sensory loss, diabetic and peripheral neuropathy.

Exclusion Criteria:

* Having had a serious lower extremity injury in the last 6 months,
* Getting a full score from the balance test,
* Having ligament rupture in the ankle.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2024-02-06 (Estimated); Primary Completion 2024-02-06 (Estimated); Study Completion 2024-07-10 (Estimated)

PRIMARY OUTCOMES:
Biodex device | 1 day
  The Biodex balance device is a specialized device used for balance training and assessment. It is designed to evaluate and improve an individual's balance, stability and proprioception. The system includes a computerized platform that provides real-time feedback and exercises for balance training. It allows assessment in the anterior and medial and posterior direction.
Y Balance Test | 1 day
  The Y Balance Test is a functional movement assessment test used to evaluate a person's dynamic balance, core strength and proprioception ability. The Y Balance Test involves reaching movements in three directions (anterior, posteromedial and posterolateral). The person stands in the center with one leg on a Y-shaped platform and reaches with the other leg in the indicated direction as far as possible while maintaining balance. .
Foot Pressure Analysis | 1 day
  These platforms measure the force applied to the sole of the foot and load distribution through electronic sensor
The Foot Posture Index | 1 day
  The Foot Posture Index is a six-criteria observational scoring system that provides a necessary measure of foot posture when the patient is standing. This system is a clinical scale for assessing the postural structure of the foot. The anatomical and biomechanical features of the foot are assessed and foot posture is classified as neutral, pronated or supinated. Its calculation consists of six different visual criteria or markers. These criteria include hindfoot position characterized by the subtalar joint, midfoot position, protrusion of the medial longitudinal arch, abduction and adduction of the forefoot, alignment of the toes, and whether the foot is supinated or pronated. Positive scores are given when pronation is observed, while negative scores are given when supination is observed
Navicular drop | 1 day
  Navicular drop test is a test used in the evaluation of ankle and lower extremity biomechanics. This test is especially used to provide information about pronation and the placement of the navicular bone. The test includes the following steps: The person stands on a flat surface with bare feet or thin socks. The sole of the feet and ankle position are observed. The ankle and foot structure is observed while the person gives a full load (stands up fully) and walks or strides to compensate for the pressure. How much the navicular bone in the center of the sole of the foot drops under load or during movement is measured.

CONTACTS AND LOCATIONS:
Locations (1):
- Bahçehir University, Istanbul, Turkey (Türkiye)